CLINICAL TRIAL: NCT00262821
Title: A Phase III, Randomized Trial of Weekly Cisplatin and Radiation Versus Cisplatin and Tirapazamine and Radiation in Stage IB2, IIA, IIIB and IVA Cervical Carcinoma Limited to the Pelvis
Brief Title: Cisplatin and Radiation Therapy With or Without Tirapazamine in Treating Patients With Cervical Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study drug no longer available resulting in lack of study drug for participants.
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NCIC Clinical Trials Group (Network); Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00591; NCI-2009-00591 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CAN-NCIC-GOG-0219; CDR0000455555; GOG-0219 (Other: Gynecologic Oncology Group); GOG-0219 (Other: CTEP); U10CA027469 (NIH); NCT00704873 (obsolete NCT alias)
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Cell Carcinoma; Cervical Squamous Cell Carcinoma; Stage IB Cervical Cancer; Stage IIA Cervical Cancer; Stage IIB Cervical Cancer; Stage III Cervical Cancer; Stage IVA Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Tirapazamine

ARMS (2):
- Arm I (cisplatin) (Active Comparator): Patients receive cisplatin IV on days 1, 8, 15, 22, 29, and 36 (weeks 1-6).
  Interventions: Drug: cisplatin
- Arm II (cisplatin, tirapazamine) (Experimental): Patients receive tirapazamine IV over 2 hours on days 1, 8, 10, 12, 15, 22, 24, 26, and 29 and cisplatin IV over 1 hour on days 1, 15, and 29.
  Interventions: Drug: cisplatin; Drug: tirapazamine

INTERVENTIONS:
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: tirapazamine — Given IV
  Other Names: SR 4233; Tirazone; WIN 59075
  Arms: Arm II (cisplatin, tirapazamine)

SUMMARY:
This randomized phase III trial is studying cisplatin, radiation therapy, and tirapazamine to see how well they work compared to cisplatin and radiation therapy in treating patients with cervical cancer. Drugs used in chemotherapy, such as cisplatin and tirapazamine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. Cisplatin and tirapazamine may make tumor cells more sensitive to radiation therapy. It is not yet known whether giving cisplatin together with radiation therapy is more effective with or without tirapazamine in treating cervical cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare the progression-free survival of patients with stage IB, IIA, IIB, IIIB, or IVA carcinoma of the cervix treated with cisplatin and radiotherapy with vs without tirapazamine.

SECONDARY OBJECTIVES:

I. Compare overall survival of patients treated with these regimens. II. Compare the toxicity of these regimens in these patients.

TERTIARY OBJECTIVES:

I. Correlate study treatment with tumor expression of carbonic anhydrase IX (CA-IX) and recurrence-free survival, overall survival, or metastasis in patients treated with these regimens.

II. Correlate expression of CA-IX, hypoxia inducible factor-1α, CD-31, thrombospondin-1, CD-105, or vascular endothelial growth factor (VEGF) in primary tumor tissue with recurrence-free survival, overall survival, or metastasis in patients treated with these regimens.

III. Correlate pre-treatment and/or post-treatment serum concentrations of angiogenic markers including angiogenin or VEGF with recurrence-free survival, overall survival, or metastasis in patients treated with these regimens.

IV. Correlate various combinations of biological markers of hypoxia and angiogenesis with recurrence-free survival, overall survival, or metastasis in patients treated with these regimens.

V. Correlate levels of individual biological markers of hypoxia or angiogenesis with clinicopathological characteristics including tumor size, histologic subtype, FIGO stage, depth of invasion, pelvic node status, site of recurrence, and hemoglobin level as well as patient, age, race and performance status in patients treated with these regimens.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are stratified according to FIGO stage of disease (IB2 vs IIA vs IIB vs IIIB vs IVA), brachytherapy method (low-dose rate vs high-dose rate), surgical staging of para-aortic nodes (yes vs no). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cisplatin IV over 30-60 minutes once weekly on days 1, 8, 15, 22, 29, and 36 (weeks 1-6). Patients also undergo external beam radiotherapy to the pelvis once daily on days 1-5, 8-12, 15-19, 22-26, and 29-33 (weeks 1-5). Patients then receive either 1 or 2 applications of low-dose rate brachytherapy in weeks 6-8 OR 5 applications of high-dose rate (HDR)* brachytherapy once weekly in weeks 4-8 and 3-5 days of parametrial boost radiotherapy** beginning after the first brachytherapy implant. Treatment continues in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive tirapazamine IV over 2 hours on days 1, 8, 10, 12, 15, 22, 24, 26, and 29 and cisplatin IV over 1 hour on days 1, 15, and 29. Patients also undergo radiotherapy and brachytherapy as in arm I. Treatment continues in the absence of disease progression or unacceptable toxicity.

NOTE: *No external beam radiotherapy is administered on the day of HDR brachytherapy. If the majority of external beam radiotherapy has been administered, HDR brachytherapy may be administered in 2 applications per week (separated by at least 72 hours) in order to complete all treatment within 8 weeks.

NOTE: ** Patients may receive a parametrial boost at the discretion of the treating radiation oncologist.

After completion of study treatment, patients are followed for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma of the uterine cervix

  * Stage IB2, IIA, IIB, IIIB, or IVA disease

    * Stage IIA tumors must be > 4 cm
  * Primary, untreated disease
* Negative, non-suspicious para-aortic nodes by lymphangiogram, CT scan, MRI, or lymphadenectomy
* Must have been adequately clinically staged
* Suitable for treatment with radical intent using concurrent chemotherapy and pelvic radiotherapy
* No disease involvement of the lower third of the vagina regardless of stage (all stage IIIA, IIIB and IVA with lower one-third involvement)
* No carcinoma of the cervical stump
* Performance status - GOG 0-3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT ≤ 3 times ULN
* Alkaline phosphatase ≤ 3 times ULN
* Creatinine ≤ ULN or calculated creatinine clearance ≥ 60mL/min
* No New York Heart Association class III-IV heart failure
* No history of myocardial infarction
* No unstable angina
* No uncontrolled hypertension
* No pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No septicemia or severe infection
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No prior hysterectomy or planned hysterectomy as part of initial cervix cancer therapy
* No prior coronary artery bypass surgery
* No prior cancer therapy that would preclude study treatment
* No concurrent angina medication
* No concurrent intensity-modulated radiotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2006-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul DiSilvestro, Principal Investigator — Gynecologic Oncology Group
Locations (282):
- United States (273):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Western Regional CCOP, Phoenix, Arizona
  - Highlands Oncology Group PA - Fayetteville, Fayetteville, Arkansas
  - Washington Regional Medical Center - Fayetteville, Fayetteville, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - East Bay Radiation Oncology Center, Castro Valley, California
  - City of Hope Medical Center, Duarte, California
  - Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Bay Area Tumor Institute CCOP, Oakland, California
  - University of California Medical Center At Irvine-Orange Campus, Orange, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Stanford University Hospitals and Clinics, Stanford, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Colorado Gynecologic Oncology Group, Aurora, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Hawaii Minority Based CCOP, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Advocate Lutheran General Hospital., Park Ridge, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University Medical Center, Indianapolis, Indiana
  - Gynecologic Oncology of Indiana, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Union Hospital of Cecil County, Elkton, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Spectrum Health-Blodgett Campus, Grand Rapids, Michigan
  - Gynecologic Oncology of West Michigan PLLC, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Providence Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Ozark Health Ventures LLC-Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Good Samaritan Hospital, Kearney, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Mountainside Hospital, Montclair, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - UMDNJ - New Jersey Medical School, Newark, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Island Gynecologic Oncology, Brightwaters, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Queens Hospital Center, Jamaica, New York
  - North Shore University Hospital, Manhasset, New York
  - North Shore-LIJ Health System CCOP, Manhasset, New York
  - Orange Regional Medical Center, Middletown, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - North Shore-LIJ Health System/Center for Advanced Medicine, New Hyde Park, New York
  - New York University Langone Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Weiler Division, The Bronx, New York
  - Good Samaritan Hospital Medical Center, West Islip, New York
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates-Midtown, Tulsa, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Salem Hospital, Salem, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Chattanooga Gynecological Oncology, Chattanooga, Tennessee
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - East Tennessee State University, Johnson City, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - American Fork Hospital, American Fork, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Fletcher Allen Health Care-Medical Center, Burlington, Vermont
  - Northern Virginia Pelvic Surgery Associates, Annandale, Virginia
  - University of Virginia, Charlottesville, Virginia
  - Bon Secours Mary Immaculate Hospital, Newport News, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Good Samaritan Community Hospital, Puyallup, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Northwest CCOP, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Tacoma General Hospital, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - Wheeling Hospital, Wheeling, West Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- Canada (9):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA-Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Health Sciences North, Greater Sudbury, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - CHUQ - Pavilion Hotel-Dieu de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

REFERENCES:
- [Derived] DiSilvestro PA, Ali S, Craighead PS, Lucci JA, Lee YC, Cohn DE, Spirtos NM, Tewari KS, Muller C, Gajewski WH, Steinhoff MM, Monk BJ. Phase III randomized trial of weekly cisplatin and irradiation versus cisplatin and tirapazamine and irradiation in stages IB2, IIA, IIB, IIIB, and IVA cervical carcinoma limited to the pelvis: a Gynecologic Oncology Group study. J Clin Oncol. 2014 Feb 10;32(5):458-64. doi: 10.1200/JCO.2013.51.4265. Epub 2014 Jan 6. PMID 24395863

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible and evaluable patients.
Groups:
- Concurrent Cisplatin and Radiation: Cisplatin, 40 mg/m2 (max = 70 mg) IV on days 1, 8, 15, 22, 29 and 36). Radiation, Pelvic (41.4-45.0 Gy / 23-25 daily fractions) brachytherapy (LDR or HDR) / boost (5.4-9.0 Gy /3-5 daily fractions) to involved parametrium
- Concurrent Cisplatin, Tirapazamine and Radiation: Cisplatin, 60 mg/m2 IV on days 1, 15 and 29; Tirapazamine,220 mg/m2 (max=385 mg) on days 1, 8, 10, 12, 15, 22, 24, 26 and 29; Radiation, Pelvic (41.4-45.0 Gy / 23-25 daily fractions) brachytherapy (LDR or HDR) / boost (5.4-9.0 Gy /3-5 daily fractions) to involved parametrium
Period: Overall Study
Arm/Group | Concurrent Cisplatin and Radiation | Concurrent Cisplatin, Tirapazamine and Radiation
Started | 198 | 204
Completed | 194 | 185
Not Completed | 4 | 19
Not completed — Ineligible - wrong stage | 0 | 3
Not completed — Ineligible - wrong cell type | 2 | 2
Not completed — Ineligible - wrong primary | 0 | 1
Not completed — Ineligible - inadequate pathology | 1 | 3
Not completed — Ineligible - elevated creatinine | 0 | 2
Not completed — Ineligible - required test not done | 1 | 4
Not completed — Inevaluable - inadequate data | 0 | 4

BASELINE CHARACTERISTICS:
Population: Eligible and evaluable patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Concurrent Cisplatin and Radiation | Concurrent Cisplatin, Tirapazamine and Radiation | Total
Number analyzed (Participants) | 194 | 185 | 379
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (11.3) | 48.4 (11.3) | 48.7 (11.3)
Age, Customized [Number; unit: participants]
  20-30 years | 7 | 10 | 17
  31-40 years | 41 | 37 | 78
  41-50 years | 65 | 61 | 126
  51-60 years | 53 | 48 | 101
  61-70 years | 20 | 23 | 43
  71-79 years | 8 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 185 | 379
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 24 | 44
  Not Hispanic or Latino | 161 | 138 | 299
  Unknown or Not Reported | 13 | 23 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 2 | 10
  Asian | 6 | 10 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 43 | 30 | 73
  White | 129 | 134 | 263
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 7 | 14
Gynecologic Oncology Group (GOG) Performance Status [Number; unit: participants] — 5-point, ordinal scale specifying patient's ability to perform activities
  participants
    0 - fully active | 147 | 141 | 288
    1 - restricted strenuous activity, ambulatory | 46 | 41 | 87
    2 - ambulatory, difficulty walking | 1 | 2 | 3
    3 - limited self-care, partly confined to bed | 0 | 1 | 1
    4 - completely disabled, no self-care | 0 | 0 | 0
Tumor Grade [Number; unit: participants] — Tumor grade was obtained from the central GOG Pathology Committee review
  participants
    1 - Well differentiated | 8 | 12 | 20
    2 - Moderately differentiated | 105 | 103 | 208
    3 - Poorly differentiated | 78 | 67 | 145
    Not graded | 3 | 3 | 6
International Federation of Gynecologic and Obstetrics (FIGO), Clinical Staging, for Cervical Carcin [Number; unit: participants] — International Federation of Gynecologic and Obstetrics (FIGO), Clinical Staging, for Cervical Carcinoma (1995). Stage IB is defined as clinical lesions confined to the cervix or pre-clinical lesions greater than stage 1A. Stage IIA is defined as the carcinoma extends beyond the cervix but has not extended on to the pelvic wall with no obvious parametrial involvement. Stage IIB has obvious parametrial involvement. Stage IIIB includes extension on to the pelvic wall and/or hydro-nephrosis or non-functioning kidney. Stage IVA is the spread of the growth to adjacent organs.
  participants
    IB | 33 | 32 | 65
    IIA | 11 | 12 | 23
    IIB | 93 | 82 | 175
    IIIB | 51 | 52 | 103
    IVA | 6 | 7 | 13
Histologic Type [Number; unit: participants] — Histologic (cell) type was obtained from the central GOG Pathology Committee review
  participants
    Squamous cell carcinoma | 164 | 158 | 322
    Adenocarcinoma, unspecified | 15 | 18 | 33
    Adenosquamous carcinoma | 11 | 5 | 16
    Other | 4 | 4 | 8
Para-aortic Lymph Node [Number; unit: participants]
  Not sampled | 25 | 33 | 58
  Sampled | 169 | 152 | 321
Brachytherapy [Number; unit: participants]
  None | 4 | 5 | 9
  Low-dose rate | 52 | 51 | 103
  High-dose rate | 138 | 129 | 267
Cooperative Group Enrollment [Number; unit: participants]
  Gynecologic Oncology Group (GOG) | 167 | 167 | 334
  National Cancer Institute of Canada (NCIC) | 24 | 17 | 41
  Other | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival - Percentage of Patients Alive and Progression Free
Description: Patients' progression status based on clinical, radiological or pathological (histological) evidence of disease after study therapy. Progression includes any death without evidence of disease progression. Progression-free Survival (PFS) is defined as time in month from study enrollment to disease progression, death or date of last contact.
Time Frame: From study entry until first disease progression, death or date of last contact, up to 6 years
Population: Eligible and evaluable patients
Measure: Number; unit: percentage of patients
Arm/Group | Concurrent Cisplatin and Radiation | Concurrent Cisplatin, Tirapazamine and Radiation
Number analyzed (Participants) | 194 | 185
percentage of patients | 64.4 | 63.0

2. Secondary Outcome: Overall Survival
Description: The observed length of life from entry into the study to death or date of last contact.
Time Frame: From study entry to death or last contact, up to 6 years
Population: Eligible and evaluable patients
Measure: Number; unit: percentage of patients alive
Arm/Group | Concurrent Cisplatin and Radiation | Concurrent Cisplatin, Tirapazamine and Radiation
Number analyzed (Participants) | 194 | 185
percentage of patients alive | 70.6 | 70.5

3. Secondary Outcome: Adverse Events (Grade 3 or Higher) During Treatment Period
Description: Number of participants with a maximum grade of 3 or higher during treatment period. Adverse events are graded and categorized using CTCAE v3.0.
Time Frame: All Adverse Events (AEs) occuring during treatment and up to 30 days after stopping the study treatment are reported
Population: All Treated Patients
Measure: Number; unit: participants
Arm/Group | Concurrent Cisplatin and Radiation | Concurrent Cisplatin, Tirapazamine and Radiation
Number analyzed (Participants) | 190 | 180
participants
  Number Participants Analyzed | 190 | 180
  Leukopenia | 51 | 53
  Thrombocytopenia | 8 | 6
  Neutropenia | 30 | 26
  Anemia | 16 | 12
  Other hematologic | 20 | 17
  Allergy/Immunology | 0 | 2
  Cardiac | 3 | 4
  Coagulation | 0 | 1
  Constitutional | 15 | 23
  Dermatologic | 0 | 17
  Gastrointestinal | 28 | 35
  Genitourinary/Renal | 4 | 4
  Hemorrhage | 5 | 5
  Infection | 14 | 14
  Metabolic | 28 | 45
  Musculoskeletal | 0 | 5
  Neuropathy | 1 | 1
  Other Neurological | 5 | 14
  Pain | 10 | 38
  Pulmonary | 3 | 6
  Vascular Disorders | 11 | 7
  Death, Not CTC Coded | 4 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported.
Description: Incidence of SAE among eligible and evaluable, treated patients.
Arm/Group | Concurrent Cisplatin and Radiation | Concurrent Cisplatin, Tirapazamine and Radiation
Serious Adverse Events (participants affected / at risk) | 42/190 | 65/180
Other Adverse Events (participants affected / at risk) | 187/190 | 179/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Concurrent Cisplatin and Radiation (N=190) | Concurrent Cisplatin, Tirapazamine and Radiation (N=180)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 0 | 1
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 0 | 1
Neutrophils (Blood and lymphatic system disorders) | 0 | 1
Platelets (Blood and lymphatic system disorders) | 0 | 1
Leukocytes (Blood and lymphatic system disorders) | 2 | 1
Lymphopenia (Blood and lymphatic system disorders) | 5 | 4
Hemoglobin (Blood and lymphatic system disorders) | 2 | 1
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 0 | 1
Ventricular Arrhythmia - Fibrillation (Cardiac disorders) | 0 | 1
Cardiac General - Other (Cardiac disorders) | 0 | 1
Fever (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 0
Death No Ctcae Term - Death Nos (General disorders) | 2 | 0
Death No Ctcae Term - Multi-Organ Failure (General disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Obstruction, Gi - Ileum (Gastrointestinal disorders) | 1 | 0
Ulcer,gi - Esophagus (Gastrointestinal disorders) | 0 | 1
Distention (Gastrointestinal disorders) | 0 | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 5
Anorexia (Gastrointestinal disorders) | 0 | 1
Dehydration (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 0 | 2
Stricture, Gi - Rectum (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 5
Hemorrhage, Gu - Vagina (Vascular disorders) | 2 | 2
Hemorrhage, Gu - Uterus (Vascular disorders) | 0 | 1
Hemorrhage, Gu - Bladder (Vascular disorders) | 0 | 1
Hemorrhage/Bleeding - Other (Vascular disorders) | 1 | 0
Liver Dysfunction (Hepatobiliary disorders) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 2 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Soft Tissue Nos (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 1 | 0
Febrile Neutropenia (Infections and infestations) | 2 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 1 | 0
Infection - Other (Infections and infestations) | 1 | 0
Inf W/Gr 3 Or 4 Anc: Bladder (Urinary) (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Pelvis Nos (Infections and infestations) | 0 | 1
Inf Unknown Anc: Rectum (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 1 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 0 | 1
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 1 | 0
Creatinine (Metabolism and nutrition disorders) | 0 | 3
Alt (Metabolism and nutrition disorders) | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
Syncope (Nervous system disorders) | 0 | 1
Mood Alteration - Depression (Nervous system disorders) | 1 | 2
Mood Alteration - Anxiety (Nervous system disorders) | 0 | 2
Cognitive Disturbance (Nervous system disorders) | 0 | 1
Pain - Other (General disorders) | 1 | 1
Pain: Pelvis (General disorders) | 0 | 2
Pain: Chest /Thorax Nos (General disorders) | 1 | 1
Pain: Back (General disorders) | 0 | 1
Pain: Abdominal Pain Nos (General disorders) | 1 | 2
Pain: Cardiac/ Heart (General disorders) | 0 | 1
Pain: Muscle (General disorders) | 0 | 1
Ards (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renal/Genitourinary - Other (Renal and urinary disorders) | 0 | 1
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Urinary Frequency (Renal and urinary disorders) | 0 | 1
Vascular - Other (Vascular disorders) | 1 | 0
Artery Injury - Aorta (Vascular disorders) | 0 | 1
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 0 | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 8 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Concurrent Cisplatin and Radiation (N=190) | Concurrent Cisplatin, Tirapazamine and Radiation (N=180)
Allergy/Immunology - Other (Immune system disorders) | 0 | 1
Allergic Reaction/Hypersensitivity (Immune system disorders) | 4 | 6
Rhinitis (Immune system disorders) | 3 | 4
Auditory/Ear - Other (Ear and labyrinth disorders) | 3 | 2
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 1 | 4
Tinnitus (Ear and labyrinth disorders) | 22 | 25
Hearing (Monitoring Program) (Ear and labyrinth disorders) | 2 | 0
Neutrophils (Blood and lymphatic system disorders) | 86 | 78
Platelets (Blood and lymphatic system disorders) | 73 | 66
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 6 | 6
Leukocytes (Blood and lymphatic system disorders) | 139 | 128
Lymphopenia (Blood and lymphatic system disorders) | 21 | 16
Hemoglobin (Blood and lymphatic system disorders) | 153 | 135
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 2 | 2
Ventricular Arrhythmia - Tachycardia (Cardiac disorders) | 1 | 1
Supraventricular Extrasystoles (Cardiac disorders) | 0 | 1
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 2 | 4
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
S/N Arrhythmia:supraventricular Nos (Cardiac disorders) | 1 | 0
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 1 | 0
Ventricular Arrhythmia - Pvcs (Cardiac disorders) | 0 | 1
Ventricular Arrhythmia - Trigeminny (Cardiac disorders) | 0 | 1
S/N Arrhythmia: Atrial Tachycardia (Cardiac disorders) | 1 | 0
Cardiac Ischemia/Infarction (Cardiac disorders) | 1 | 1
Hypertension (Cardiac disorders) | 10 | 5
Cardiac General - Other (Cardiac disorders) | 1 | 0
Cardiac Troponin T (Ctnt) (Cardiac disorders) | 0 | 1
Hypotension (Cardiac disorders) | 2 | 5
Inr (Vascular disorders) | 0 | 1
Constitutional Symptoms - Other (General disorders) | 2 | 2
Sweating (General disorders) | 6 | 3
Weight Gain (General disorders) | 1 | 1
Fever (General disorders) | 12 | 10
Weight Loss (General disorders) | 35 | 43
Rigors/Chills (General disorders) | 2 | 3
Fatigue (General disorders) | 140 | 134
Insomnia (General disorders) | 22 | 21
Nail Changes (Skin and subcutaneous tissue disorders) | 4 | 0
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 2 | 3
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 12 | 14
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 3
Dermatitis - Chemoradiation (Skin and subcutaneous tissue disorders) | 1 | 0
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 0 | 1
Bruising (Skin and subcutaneous tissue disorders) | 3 | 2
Acne (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 12 | 43
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 6
Decubitus (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis - Radiation (Skin and subcutaneous tissue disorders) | 26 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 13
Burn (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 5 | 7
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 8
Hot Flashes (Endocrine disorders) | 21 | 12
Enteritis (Gastrointestinal disorders) | 1 | 0
Obstruction, Gi - Ileum (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 2 | 1
Flatulence (Gastrointestinal disorders) | 3 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 4 | 3
Hemorrhoids (Gastrointestinal disorders) | 7 | 2
Heartburn (Gastrointestinal disorders) | 19 | 13
Perforation, Gi - Rectum (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 3
Distention (Gastrointestinal disorders) | 1 | 1
Taste Alteration (Gastrointestinal disorders) | 28 | 27
Incontinence, Anal (Gastrointestinal disorders) | 1 | 2
Dry Mouth (Gastrointestinal disorders) | 4 | 8
Mucositis (Functional/Sympt) - Rectum (Gastrointestinal disorders) | 1 | 0
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 3 | 9
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1
Necrosis, Gi - Rectum (Gastrointestinal disorders) | 0 | 1
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 8 | 10
Vomiting (Gastrointestinal disorders) | 75 | 107
Anorexia (Gastrointestinal disorders) | 59 | 60
Dehydration (Gastrointestinal disorders) | 7 | 19
Constipation (Gastrointestinal disorders) | 50 | 47
Nausea (Gastrointestinal disorders) | 127 | 134
Gastrointestinal - Other (Gastrointestinal disorders) | 6 | 3
Diarrhea (Gastrointestinal disorders) | 119 | 112
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 3 | 1
Hemorrhage, Gu - Vagina (Vascular disorders) | 39 | 28
Hemorrhage, Gi - Rectum (Vascular disorders) | 2 | 3
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 1 | 1
Hematoma (Vascular disorders) | 1 | 0
Hemorrhage, Gi - Anus (Vascular disorders) | 1 | 0
Hemorrhage, Gu - Uterus (Vascular disorders) | 0 | 1
Hemorrhage, Gi - Oral Cavity (Vascular disorders) | 0 | 1
Hemorrhage, Gu - Kidney (Vascular disorders) | 0 | 1
Hemorrhage, Gu - Bladder (Vascular disorders) | 2 | 1
Petechiae (Vascular disorders) | 1 | 0
Hemorrhage/Bleeding - Other (Vascular disorders) | 1 | 0
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Artery (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Vulva (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Cervix (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 1 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Oral Cavity-Gums (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 2 | 0
Febrile Neutropenia (Infections and infestations) | 0 | 2
Inf Unknown Anc: Nerve-Peripheral (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Colon (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 10 | 15
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 1 | 0
Infection - Other (Infections and infestations) | 0 | 3
Inf W/Gr 3 Or 4 Anc: Bladder (Urinary) (Infections and infestations) | 1 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Nerve-Peripheral (Infections and infestations) | 1 | 0
Inf W/Gr 3 Or 4 Anc: Oral Cavity-Gums (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Pharynx (Infections and infestations) | 0 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Vagina (Infections and infestations) | 2 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Pelvis Nos (Infections and infestations) | 1 | 0
Inf Unknown Anc: Bronchus (Infections and infestations) | 1 | 0
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 4 | 0
Inf Unknown Anc: Bladder (Urinary) (Infections and infestations) | 1 | 1
Inf Unknown Anc: Rectum (Infections and infestations) | 1 | 0
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Anal/Perianal (Infections and infestations) | 0 | 1
Inf W/Gr 3 Or 4 Anc: Lung (Pneumonia) (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 2 | 6
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 3 | 0
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 0 | 2
Edema: Limb (Blood and lymphatic system disorders) | 12 | 13
Edema: Head And Neck (Blood and lymphatic system disorders) | 0 | 2
Ast (Metabolism and nutrition disorders) | 4 | 20
Gfr (Metabolism and nutrition disorders) | 3 | 4
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 4 | 8
Proteinuria (Metabolism and nutrition disorders) | 1 | 0
Creatinine (Metabolism and nutrition disorders) | 22 | 21
Hypoalbuminemia (Metabolism and nutrition disorders) | 22 | 37
Ggt (Metabolism and nutrition disorders) | 5 | 7
Alt (Metabolism and nutrition disorders) | 6 | 27
Alkaline Phosphatase (Metabolism and nutrition disorders) | 8 | 17
Bilirubin (Metabolism and nutrition disorders) | 5 | 5
Lipase (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 4 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 6
Hyponatremia (Metabolism and nutrition disorders) | 40 | 46
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 4 | 3
Amylase (Metabolism and nutrition disorders) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 2 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 32 | 37
Hyperkalemia (Metabolism and nutrition disorders) | 7 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 46 | 61
Hypokalemia (Metabolism and nutrition disorders) | 40 | 61
Hypoglycemia (Metabolism and nutrition disorders) | 8 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 52 | 51
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 4 | 14
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint-Function (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 10 | 6
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 2 | 1
Neuropathy,cranial - Cn X Motor-Palate (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 4
Involuntary Movement (Nervous system disorders) | 1 | 0
Psychosis (Nervous system disorders) | 1 | 0
Neurology - Other (Nervous system disorders) | 3 | 2
Encephalopathy (Nervous system disorders) | 0 | 1
Mood Alteration - Depression (Nervous system disorders) | 18 | 12
Mood Alteration - Anxiety (Nervous system disorders) | 15 | 18
Mood Alteration - Agitation (Nervous system disorders) | 0 | 3
Tremor (Nervous system disorders) | 2 | 2
Personality (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Confusion (Nervous system disorders) | 2 | 4
Memory Impairment (Nervous system disorders) | 2 | 3
Dizziness (Nervous system disorders) | 20 | 22
Neuropathy,cranial - Cn I Smell (Nervous system disorders) | 1 | 2
Neuropathy-Sensory (Nervous system disorders) | 31 | 30
Neuropathy-Motor (Nervous system disorders) | 1 | 12
Ocular/Visual - Other (Eye disorders) | 0 | 3
Dry Eye (Eye disorders) | 1 | 2
Photophobia (Eye disorders) | 0 | 1
Flashing Lights/Floaters (Eye disorders) | 1 | 5
Diplopia (Eye disorders) | 2 | 0
Blurred Vision (Eye disorders) | 6 | 11
Pain - Other (General disorders) | 9 | 12
Pain: Urethra (General disorders) | 6 | 10
Pain: Perineum (General disorders) | 0 | 1
Pain: Pelvis (General disorders) | 27 | 28
Pain: Vagina (General disorders) | 11 | 6
Pain: Uterus (General disorders) | 1 | 0
Pain: Chest /Thorax Nos (General disorders) | 0 | 6
Pain: Chest Wall (General disorders) | 3 | 0
Pain: Throat/Pharynx/Larynx (General disorders) | 2 | 1
Pain: Head/Headache (General disorders) | 25 | 15
Pain: Neck (General disorders) | 2 | 0
Pain: Extremity-Limb (General disorders) | 13 | 28
Pain: Buttock (General disorders) | 1 | 2
Pain: Back (General disorders) | 23 | 21
Pain: Joint (General disorders) | 6 | 2
Pain: Bone (General disorders) | 4 | 2
Pain: Kidney (General disorders) | 0 | 2
Pain: Bladder (General disorders) | 9 | 7
Pain: Pain Nos (General disorders) | 5 | 1
Pain: Stomach (General disorders) | 3 | 3
Pain: Rectum (General disorders) | 5 | 7
Pain: Peritoneum (General disorders) | 1 | 0
Pain: Oral Cavity (General disorders) | 1 | 0
Pain: Esophagus (General disorders) | 0 | 1
Pain: Dental/Teeth/Peridontal (General disorders) | 0 | 1
Pain: Abdominal Pain Nos (General disorders) | 52 | 36
Pain: Cardiac/ Heart (General disorders) | 1 | 1
Pain: Tumor (General disorders) | 3 | 1
Pain: Muscle (General disorders) | 12 | 48
Pain: Anus (General disorders) | 1 | 1
Pain: Neuralgia (General disorders) | 1 | 0
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 | 15
Renal/Genitourinary - Other (Renal and urinary disorders) | 3 | 2
Stricture, Anastomotic, Gu - Urethra (Renal and urinary disorders) | 1 | 0
Stricture, Anastomotic, Gu - Ureter (Renal and urinary disorders) | 1 | 0
Leak, Gu - Vagina (Renal and urinary disorders) | 1 | 0
Cystitis (Renal and urinary disorders) | 27 | 17
Urinary Color Change (Renal and urinary disorders) | 1 | 2
Urinary Retention (Renal and urinary disorders) | 1 | 4
Obstruction, Gu - Urethra (Renal and urinary disorders) | 1 | 0
Obstruction, Gu - Ureter (Renal and urinary disorders) | 3 | 1
Obstruction, Gu - Bladder (Renal and urinary disorders) | 0 | 1
Incontinence, Urinary (Renal and urinary disorders) | 6 | 4
Fistula, Gu - Vagina (Renal and urinary disorders) | 2 | 0
Bladder Spasm (Renal and urinary disorders) | 12 | 8
Renal Failure (Renal and urinary disorders) | 0 | 1
Urinary Frequency (Renal and urinary disorders) | 28 | 13
Vaginal Dryness (Reproductive system and breast disorders) | 0 | 2
Sexual/Reproductive Function: Other (Reproductive system and breast disorders) | 1 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 30 | 14
Syndromes - Other (General disorders) | 1 | 0
Vascular - Other (Vascular disorders) | 1 | 0
Vein Injury - Extremity-Upper (Vascular disorders) | 1 | 0
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 0 | 2
Thrombosis/Thrombus/Embolism (Vascular disorders) | 3 | 2
Phlebitis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Premature closure due to lack of study drug leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less